CLINICAL TRIAL: NCT05614167
Title: Relationship Between Isometric Muscle Strength and Gross Motor Function in Children With Unilateral Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Omnya Samy Abdallah Ghoneim, Lecturer, Department of Physical Therapy for Pediatrics and Pediatric Surgery, Faculty of Physical Therapy, Badr University in Cairo, Egypt., Badr University
Other Study IDs: Omnya3
Record Dates: First submitted 2022-11-05; First posted 2022-11-14 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Hemiplegia; Cerebral Palsy
Keywords: Hemiplegia; Cerebral Palsy; muscle stength; gmfm
MeSH Terms: conditions — Hemiplegia; Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: correlation — A total of 97 children with CP between the ages of six and 12 years participated in the study. Muscle strength was measured with a handheld dynamometer. Motor function in children with CP was classified with the Gross Motor Function Classification System (GMFCS), graded with the Gross Motor Function Measure (GMFM)

SUMMARY:
Muscle strength can be defined as the ability of skeletal muscle to develop force for the purpose of providing stability and mobility within the musculoskeletal system, so that functional movement can take place.

DETAILED DESCRIPTION:
Cerebral palsy describes a group of disorders of the development of movement and posture, causing activity limitation, that are attributed to non-progressive disturbances that occurred in the developing fatal or infant brain. The motor disorders of cerebral palsy are often accompanied by disturbances of sensation, cognition, communication, perception, and/or behaviour, and/or by a seizure disorder

The development and changes in motor function, both natural and with therapy, can be assessed using the Gross Motor Function Measure (GMFM) created for children with CP

ELIGIBILITY:
Inclusion Criteria:

1. Their age between 6 and 12 years old.
2. Grade 1and 2 according to the Modified Ashworth scale (RW and Smith, 1987).
3. They could walk with limitation or holding on according to GMFCS (level I, II) (Palisano et al., 1997).
4. They were able to understand and follow verbal instructions.

Exclusion Criteria:

1. Children with any visual or auditory problems.
2. Children with any surgical interference in the lower limb.
3. Children with any structural deformities in joints and bones of lower limbs.
4. Children with any special medications affecting muscle functions (anti-spastic drugs).
5. Children who suffer from other diseases or associated disorders that interfered with physical activity.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Muscle weakness was found in children with CP, increasing with severity of gross motor function, approximately 50% of the predicted muscle strength was needed to be able to walk without aids.
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-02-12 (Actual)

PRIMARY OUTCOMES:
Gross motor function measure | 3 months
  standing and walking domain
Isometric muscle strength | 3 months
  a handheld dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Omnya samy, PHD, Principal Investigator — lecturer
Locations (1):
- Badr University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
private